CLINICAL TRIAL: NCT03004911
Title: Development of a Mobile Application to Promote Self-care in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 274/14
Record Dates: First submitted 2016-12-21; First posted 2016-12-29 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2016-12

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; mobile application; self-care; quality of life
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile application (Experimental)
  Interventions: Device: ProFibro (Mobile application)
- Paper booklet (Active Comparator)
  Interventions: Device: Paper booklet

INTERVENTIONS:
Device: ProFibro (Mobile application) — ProFibro, a mobile Android application in Brazilian Portuguese to promote self-care in patients with fibromyalgia
  Arms: Mobile application
Device: Paper booklet — A 64-page booklet with content similar to the mobile application
  Arms: Paper booklet

SUMMARY:
The purpose of this study is to test the efficacy of a mobile application named ProFibro to promote self-care, and improve symptoms and health-related quality of life in Brazilian patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of fibromyalgia, according to the 2010 American College of Rheumatology diagnostic criteria
* smartphone user
* complete primary education

Exclusion Criteria:

* being in physical therapy treatment for fibromyalgia or having been treated in the last 3 months
* diagnosis of other chronic pain conditions (neuropathies, rheumatoid arthritis, osteoarthritis, spinal stenosis or cancer)
* severe mental disorders (schizophrenia, psychosis, bipolar affective disorder, severe depression)
* moderate or severe intellectual disability
* hearing or visual impairment

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan LK Yuan, MSc, Principal Investigator — Rehabilitation Sciences PhD program of the School of Medicine of the University of Sao Paulo; Amelia P Marques, PhD, Study Chair — Department of Physical Therapy, Speech Therapy and Occupational Therapy of the School of Medicine of the University of Sao Paulo
Locations (1):
- Department of Physical Therapy, Speech Therapy and Occupational Therapy of the School of Medicine of the University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paiva ES, Heymann RE, Rezende MC, Helfenstein M Jr, Martinez JE, Provenza JR, Ranzolin A, de Assis MR, Pasqualin VD, Bennett RM. A Brazilian Portuguese version of the Revised Fibromyalgia Impact Questionnaire (FIQR): a validation study. Clin Rheumatol. 2013 Aug;32(8):1199-206. doi: 10.1007/s10067-013-2259-6. Epub 2013 Apr 21. PMID 23604595
- [Background] Bennett RM, Bushmakin AG, Cappelleri JC, Zlateva G, Sadosky AB. Minimal clinically important difference in the fibromyalgia impact questionnaire. J Rheumatol. 2009 Jun;36(6):1304-11. doi: 10.3899/jrheum.081090. Epub 2009 Apr 15. PMID 19369473
- [Background] Altman DG, Bland JM. How to randomise. BMJ. 1999 Sep 11;319(7211):703-4. doi: 10.1136/bmj.319.7211.703. No abstract available. PMID 10480833
- [Background] Henriksson C, Carlberg U, Kjallman M, Lundberg G, Henriksson KG. Evaluation of four outpatient educational programmes for patients with longstanding fibromyalgia. J Rehabil Med. 2004 Sep;36(5):211-9. doi: 10.1080/16501970410027494. PMID 15626161
- [Background] Nam S, Tin D, Bain L, Thorne JC, Ginsburg L. Clinical utility of the Hospital Anxiety and Depression Scale (HADS) for an outpatient fibromyalgia education program. Clin Rheumatol. 2014 May;33(5):685-92. doi: 10.1007/s10067-013-2377-1. Epub 2013 Sep 1. PMID 23995734
- [Background] Bennett RM, Friend R, Jones KD, Ward R, Han BK, Ross RL. The Revised Fibromyalgia Impact Questionnaire (FIQR): validation and psychometric properties. Arthritis Res Ther. 2009;11(4):R120. doi: 10.1186/ar2783. Epub 2009 Aug 10. PMID 19664287
- [Background] Bennett R. The Fibromyalgia Impact Questionnaire (FIQ): a review of its development, current version, operating characteristics and uses. Clin Exp Rheumatol. 2005 Sep-Oct;23(5 Suppl 39):S154-62. PMID 16273800
- [Background] Marques AP, Assumpcao A, Matsutani LA, Pereira CA, Lage L. Pain in fibromyalgia and discrimination power of the instruments: Visual Analog Scale, Dolorimetry and the McGill Pain Questionnaire. Acta Reumatol Port. 2008 Jul-Sep;33(3):345-51. PMID 18846013
- [Background] Sousa VD, Zauszniewski JA, Bergquist-Beringer S, Musil CM, Neese JB, Jaber AF. Reliability, validity and factor structure of the Appraisal of Self-Care Agency Scale-Revised (ASAS-R). J Eval Clin Pract. 2010 Dec;16(6):1031-40. doi: 10.1111/j.1365-2753.2009.01242.x. PMID 20626539
- [Background] Damasio BF, Koller SH. The Appraisal of Self-Care Agency Scale - Revised (ASAS-R): adaptation and construct validity in the Brazilian context. Cad Saude Publica. 2013 Oct;29(10):2071-82. doi: 10.1590/0102-311x00165312. PMID 24127101
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- See also: The website briefly explains the stages of the development of ProFibro, the main functions of the application and the test of its efficacy. — https://profibro2018.wordpress.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Mobile Application: The use of ProFibro mobile application for six weeks
- Paper Booklet: The use of a 64-page booklet (with content similar to the mobile application) for six weeks
Period: Overall Study
Arm/Group | Mobile Application | Paper Booklet
Started | 20 | 20
Completed | 19 | 17
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Mobile Application: The use of ProFibro app for 6 weeks
- Paper Booklet: The use of the booklet for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Mobile Application | Paper Booklet | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (8.4) | 42.1 (11.8) | 42.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 20 | 20 | 40
Health-related Quality of Life Assessed With the Revised Fibromyalgia Impact Questionnaire [Mean (Standard Deviation); unit: score on a scale] — Minimum value: 0. Maximum value: 100. Higher scores mean worse outcome.
  score on a scale | 62.6 (16.8) | 65.4 (18) | 64 (17.3)
Number of Painful Areas Assessed With the Widespread Pain Index [Mean (Standard Deviation); unit: number of painful areas] — Minimum value: 0. Maximum value: 19.
  number of painful areas | 13.6 (4) | 13.6 (3.7) | 13.6 (3.8)
Pain Assessed With the Visual Analogue Scale [Mean (Standard Deviation); unit: score on a scale] — Minimum value: 0. Maximum value: 10. Higher scores mean worse outcome.
  score on a scale | 5.9 (2.2) | 5.7 (2.2) | 5.8 (2.2)
Severity of Symptoms Assessed With the Symptom Severity Scale [Mean (Standard Deviation); unit: score on a scale] — Minimum value: 0. Maximum value: 12. Higher scores mean worse outcome.
  score on a scale | 9.4 (1.5) | 9.2 (1.9) | 9.3 (1.7)
Self-care Agency Assessed With the Appraisal of Self-Care Agency Scale - Revised [Mean (Standard Deviation); unit: score on a scale] — Minimum value: 15. Maximum value: 75. Higher scores mean better outcome.
  score on a scale | 51.9 (9.7) | 53.5 (11) | 52.7 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: Health-related Quality of Life Assessed With the Revised Fibromyalgia Impact Questionnaire
Description: Minimum value: 0. Maximum value: 100. Higher scores mean worse outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Application | Paper Booklet
Number analyzed (Participants) | 20 | 20
score on a scale | 53.7 (17.1) | 55.5 (18.2)
Statistical Analysis 1: Comparison: Mobile Application vs Paper Booklet; Test type: Superiority; p = 0.740, t-test, 2 sided

2. Secondary Outcome: Number of Painful Areas Assessed With the Widespread Pain Index
Description: Minimum value: 0. Maximum value: 19.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: number of painful areas
Arm/Group | Mobile Application | Paper Booklet
Number analyzed (Participants) | 20 | 20
number of painful areas | 12.5 (4.6) | 12.3 (4.5)
Statistical Analysis 1: Comparison: Mobile Application vs Paper Booklet; Test type: Superiority; p = 0.890, t-test, 2 sided

3. Secondary Outcome: Pain Assessed With the Visual Analogue Scale
Description: Minimum value: 0. Maximum value: 10. Higher scores mean worse outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Application | Paper Booklet
Number analyzed (Participants) | 20 | 20
score on a scale | 5.1 (2.6) | 5.3 (2.3)
Statistical Analysis 1: Comparison: Mobile Application vs Paper Booklet; Test type: Superiority; p = 0.747, t-test, 2 sided

4. Secondary Outcome: Severity of Symptoms Assessed With the Symptom Severity Scale
Description: Minimum value: 0. Maximum value: 12. Higher scores mean worse outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Application | Paper Booklet
Number analyzed (Participants) | 20 | 20
score on a scale | 7.6 (2.9) | 7.6 (2.4)
Statistical Analysis 1: Comparison: Mobile Application vs Paper Booklet; Test type: Superiority; p = 1.000, t-test, 2 sided

5. Secondary Outcome: Self-care Agency Assessed With the Appraisal of Self-Care Agency Scale - Revised
Description: Minimum value: 15. Maximum value: 75. Higher scores mean better outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Application | Paper Booklet
Number analyzed (Participants) | 20 | 20
score on a scale | 56.8 (10.2) | 54.3 (11)
Statistical Analysis 1: Comparison: Mobile Application vs Paper Booklet; Test type: Superiority; p = 0.459, t-test, 2 sided

6. Secondary Outcome: Adherence to Mobile Application Assessed by Number of Clicks on the App Functions
Description: Number of clicks on the app functions
Time Frame: 6 weeks
Measure: Median (Full Range); unit: Clicks on app functions
Arm/Group | Mobile Application
Number analyzed (Participants) | 20
Clicks on app functions | 106 [12 to 237]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Mobile Application | Paper Booklet
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT03004911/Prot_SAP_000.pdf